CLINICAL TRIAL: NCT03450356
Title: The German Version of the Awareness of Social Inference Test: Development of a Short and Sensitive Version for Use in Clinical Populations
Brief Title: The German Version of the Awareness of Social Inference Test
Acronym: TASIT
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01193; me15Sollberger
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Social Cognition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Goal of the current project is the development of a German-language test battery for a realistic investigation of core areas of social issues Cognition (emotion, perspective taking). This test battery should be used in the investigation of patients with neuropsychological disorders. Investigators plan to establish a German-version of the TASIT that is more sensitive and shorter in administration than the original TASIT.

ELIGIBILITY:
Inclusion Criteria:

* from the age of 35,
* at least 7 years of education
* understand German or Swiss German
* Subjective statement of good health
* Signed consent

Exclusion Criteria:

* Montreal Cognitive Assessment (MoCA) value below the fifth percentile of subjectively cognitive healthy persons
* signs of depressive mood (Geriatric Depression Scale (GDS) score ≥ 5 points or Beck Depression Inventory (BDI) ≥ 10 points)
* Severe sensory deficits with potentially negative influence test results
* Severe motor deficits with potentially negative influence test results
* Systemic diseases or brain diseases with potentially negative Influence on test results
* St. n. Traumatic brain injury (with unconsciousness of at least 30 minutes)
* Severe pain with potentially negative influence on the test results
* Psychiatric problems like alcohol dependence syndrome or Schizophrenia according to Diagnostic and Statistical Manual (DSM)®-5
* Regular use of drugs with potentially negative Influence on the test results with the exception of taking Benzodiazepines at night
* general anesthesia less than 3 months ago

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Accuracy rate in emotion perception and perception of beliefs and intentions | 60 minutes
  The proportion of top scorers for any question - i.e. the proportion of participants who reach the full score of a specific scene. This proportion will be estimated for each scene and intensity separately with 95% confidence interval.
Accuracy rate in perception of beliefs | 60 minutes
  The proportion of top scorers for any question - i.e. the proportion of participants who reach the full score of a specific scene. This proportion will be estimated for each scene and intensity separately with 95% confidence interval.
Accuracy rate in perception of intentions | 60 minutes
  The proportion of top scorers for any question - i.e. the proportion of participants who reach the full score of a specific scene. This proportion will be estimated for each scene and intensity separately with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sollberger, PD Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland